CLINICAL TRIAL: NCT00340015
Title: NCI-AARP Diet and Health Study
Brief Title: A Prospective Study of Diet and Cancer in Members of the American Association of Retired Persons
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995025; OH95-C-N025
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Death; Cancer
Keywords: Cancer; Mortality; Lifestyle Factors; Nutrition; Prospective Cohort; Natural History
MeSH Terms: conditions — Death; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- AARP: Members of the AARP, aged 50-71 years, and who resided in one of six states

SUMMARY:
This is a prospective cohort study of diet and cancer in relation to several major cancers, especially breast, prostate, and colorectal malignancies. The cohort comprises 50-69 year-old male and female members of the American Association of Retired Persons (AARP). In 1995-6 we mailed baseline questionnaires to 3.5 million AARP members. Over 615,000 AARP members responded, with over 540,000 providing adequate dietary data. Preliminary analysis indicates that the cohort, both men and women, has the desired wide distributions of percent calories from fat, dietary fiber, fruits and vegetables, and red meat. Approximately 330,000 of the initial respondents (with satisfactory data) returned a second questionnaire containing questions on exposures not assessed in the first instrument.

In terms of field activities, the study has been relatively quiescent over the past year. At the end of the five-year period of observation, we will mail to cohort members a brief follow-up questionnaire primarily targeted to endpoint assessment. (Because of cancer registry lag-time, we do not expect to mail this questionnaire until early 2002.) Follow-up will be largely passive, through established state registries. The initial questionnaire mailing will be to AARP members in those states selected on the basis of having registries with adequate coverage and quality. We will use active follow-up, with record retrieval, for the small percentage of cohort members who have moved out of the cancer registry areas. The buccal cell collection pilot study has been completed; over 50% of those pilot study partricipants who had completed the baseline and risk factor questionnaires returned buccal cell speciments. Preliminary data from a pilot study of the end point ascertainment procedure indicate that cohort incidence rates for major cancers, determined from registry data, are consistent with SEER rates.

DETAILED DESCRIPTION:
This is a prospective cohort study to investigate relations among diet, lifestyle and cancer. The cohort comprises 50-69 year-old male and female members of the American Association of Retired Persons (AARP). In 1995-96 we mailed baseline questionnaires to 3.5 million AARP members. Over 615,000 AARP members responded, with over 540,000 providing adequate dietary data. Preliminary analysis indicates that the cohort, both men and women, has the desired wide distributions of percent calories from fat, dietary fiber, fruits and vegetables, and red meat. Approximately 330,000 of the initial respondents (with satisfactory data) returned a second questionnaire containing questions on exposures not assessed in the first instrument. In 2004-2006 we mailed a follow-up questionnaire to all living participants to assess non-cancer endpoints and lifestyle factors.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients participating will be selected from the American Association of Retired Persons age 50-69 living in one of the following state and metropolitan areas: California (minus Los Angeles county), Florida, Pennsylvania, New Jersey, Louisiana, North Carolina, Detroit, and Atlanta.

Ages: 50 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Members of the AARP (formally the American Association of Retired Persons), aged 50-71 years, and who resided in one of six states (California, Florida, Pennsylvania, New Jersey, North Carolina, and Louisiana) or in two metropolitan areas (Atlanta, Georgia and Detroit, Michigan) in 1995-1996.
Sampling Method: Non-Probability Sample
Enrollment: 566401 (Actual)
Dates: Start 1995-10-24 (Actual); Primary Completion 2015-02-25 (Actual); Study Completion 2015-02-25 (Actual)

PRIMARY OUTCOMES:
Incident Cancer | 12/31/2030
  All cancers
All cause and disease specific mortality | 12/31/2030
  All cause and disease specific mortality
Chronic diseases | 12/31/2030
  Chronic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Sinha, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Zhuang P, Wu F, Mao L, Zhu F, Zhang Y, Chen X, Jiao J, Zhang Y. Egg and cholesterol consumption and mortality from cardiovascular and different causes in the United States: A population-based cohort study. PLoS Med. 2021 Feb 9;18(2):e1003508. doi: 10.1371/journal.pmed.1003508. eCollection 2021 Feb. PMID 33561122
- [Derived] Willis EA, Huang WY, Saint-Maurice PF, Leitzmann MF, Salerno EA, Matthews CE, Berndt SI. Increased frequency of intentional weight loss associated with reduced mortality: a prospective cohort analysis. BMC Med. 2020 Sep 17;18(1):248. doi: 10.1186/s12916-020-01716-5. PMID 32938465
- [Derived] Zhuang P, Zhang Y, He W, Chen X, Chen J, He L, Mao L, Wu F, Jiao J. Dietary Fats in Relation to Total and Cause-Specific Mortality in a Prospective Cohort of 521 120 Individuals With 16 Years of Follow-Up. Circ Res. 2019 Mar;124(5):757-768. doi: 10.1161/CIRCRESAHA.118.314038. PMID 30636521
- [Derived] Hashemian M, Murphy G, Etemadi A, Dawsey SM, Liao LM, Abnet CC. Nut and peanut butter consumption and the risk of esophageal and gastric cancer subtypes. Am J Clin Nutr. 2017 Sep;106(3):858-864. doi: 10.3945/ajcn.117.159467. Epub 2017 Aug 2. PMID 28768652
- [Derived] Keadle SK, Arem H, Moore SC, Sampson JN, Matthews CE. Impact of changes in television viewing time and physical activity on longevity: a prospective cohort study. Int J Behav Nutr Phys Act. 2015 Dec 18;12:156. doi: 10.1186/s12966-015-0315-0. PMID 26678502
- [Derived] Xu M, Huang T, Lee AW, Qi L, Cho S. Ready-to-Eat Cereal Consumption with Total and Cause-Specific Mortality: Prospective Analysis of 367,442 Individuals. J Am Coll Nutr. 2016;35(3):217-23. doi: 10.1080/07315724.2014.971193. Epub 2015 Nov 23. PMID 26595440
- [Derived] Keadle SK, Moore SC, Sampson JN, Xiao Q, Albanes D, Matthews CE. Causes of Death Associated With Prolonged TV Viewing: NIH-AARP Diet and Health Study. Am J Prev Med. 2015 Dec;49(6):811-21. doi: 10.1016/j.amepre.2015.05.023. Epub 2015 Jul 26. PMID 26215832
- [Derived] Kabat GC, Matthews CE, Kamensky V, Hollenbeck AR, Rohan TE. Adherence to cancer prevention guidelines and cancer incidence, cancer mortality, and total mortality: a prospective cohort study. Am J Clin Nutr. 2015 Mar;101(3):558-69. doi: 10.3945/ajcn.114.094854. Epub 2015 Jan 7. PMID 25733641
- [Derived] Matthews CE, Moore SC, Sampson J, Blair A, Xiao Q, Keadle SK, Hollenbeck A, Park Y. Mortality Benefits for Replacing Sitting Time with Different Physical Activities. Med Sci Sports Exerc. 2015 Sep;47(9):1833-40. doi: 10.1249/MSS.0000000000000621. PMID 25628179
- [Derived] Jiao L, Stolzenberg-Solomon R, Zimmerman TP, Duan Z, Chen L, Kahle L, Risch A, Subar AF, Cross AJ, Hollenbeck A, Vlassara H, Striker G, Sinha R. Dietary consumption of advanced glycation end products and pancreatic cancer in the prospective NIH-AARP Diet and Health Study. Am J Clin Nutr. 2015 Jan;101(1):126-34. doi: 10.3945/ajcn.114.098061. Epub 2014 Nov 19. PMID 25527756
- [Derived] Tasevska N, Park Y, Jiao L, Hollenbeck A, Subar AF, Potischman N. Sugars and risk of mortality in the NIH-AARP Diet and Health Study. Am J Clin Nutr. 2014 May;99(5):1077-88. doi: 10.3945/ajcn.113.069369. Epub 2014 Feb 19. PMID 24552754
- [Derived] Li WQ, Park Y, Wu JW, Goldstein AM, Taylor PR, Hollenbeck AR, Freedman ND, Abnet CC. Index-based dietary patterns and risk of head and neck cancer in a large prospective study. Am J Clin Nutr. 2014 Mar;99(3):559-66. doi: 10.3945/ajcn.113.073163. Epub 2014 Jan 8. PMID 24401718
- [Derived] Daniel CR, Park Y, Chow WH, Graubard BI, Hollenbeck AR, Sinha R. Intake of fiber and fiber-rich plant foods is associated with a lower risk of renal cell carcinoma in a large US cohort. Am J Clin Nutr. 2013 May;97(5):1036-43. doi: 10.3945/ajcn.112.045351. Epub 2013 Mar 20. PMID 23515007
- [Derived] Sinha R, Cross AJ, Daniel CR, Graubard BI, Wu JW, Hollenbeck AR, Gunter MJ, Park Y, Freedman ND. Caffeinated and decaffeinated coffee and tea intakes and risk of colorectal cancer in a large prospective study. Am J Clin Nutr. 2012 Aug;96(2):374-81. doi: 10.3945/ajcn.111.031328. Epub 2012 Jun 13. PMID 22695871
- [Derived] Daniel CR, Sinha R, Park Y, Graubard BI, Hollenbeck AR, Morton LM, Cross AJ. Meat intake is not associated with risk of non-Hodgkin lymphoma in a large prospective cohort of U.S. men and women. J Nutr. 2012 Jun;142(6):1074-80. doi: 10.3945/jn.112.158113. Epub 2012 Apr 25. PMID 22535761
- [Derived] Matthews CE, George SM, Moore SC, Bowles HR, Blair A, Park Y, Troiano RP, Hollenbeck A, Schatzkin A. Amount of time spent in sedentary behaviors and cause-specific mortality in US adults. Am J Clin Nutr. 2012 Feb;95(2):437-45. doi: 10.3945/ajcn.111.019620. Epub 2012 Jan 4. PMID 22218159
- [Derived] Daniel CR, Cross AJ, Graubard BI, Park Y, Ward MH, Rothman N, Hollenbeck AR, Chow WH, Sinha R. Large prospective investigation of meat intake, related mutagens, and risk of renal cell carcinoma. Am J Clin Nutr. 2012 Jan;95(1):155-62. doi: 10.3945/ajcn.111.019364. Epub 2011 Dec 14. PMID 22170360